CLINICAL TRIAL: NCT01009268
Title: The Effect of a Pre- and Postoperative Orthogeriatric Service. A Randomised, Controlled Trial
Brief Title: The Effect of a Pre- and Postoperative Orthogeriatric Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1361
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Dementia; Delirium
MeSH Terms: conditions — Dementia; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Orthogeriatric intervention — The intervention group will be transferred as soon as possible to the orthogeriatric ward, stabilised there preoperatively, and transferred back to the same ward postoperatively for further treatment and rehabilitation, while the control group will be treated in a traditional orthopaedic ward. Operative and anaesthesiologic procedures will be the same in the two groups.Clinical routines for the orthogeriatric service has been developed during the pilot phase in 2008 and 2009, and are documented in the electronic library of clinical handbooks at Department of Geriatric Medicine.

SUMMARY:
The investigators' aim is to assess the effect of a model of preoperative as well as early postoperative care, treatment and rehabilitation in a dedicated orthogeriatric ward in a single-blind randomised study.

The investigators' main hypothesis is that an orthogeriatric service may improve long-time cognitive outcome.

DETAILED DESCRIPTION:
The study will be carried out in close cooperation between the Orthopaedic Centre and the Department of Geriatric Medicine. The patients will be randomized in the Emergency Department in accordance with procedures already established for a recently finished trial. The intervention group will be transferred as soon as possible to the orthogeriatric ward, stabilised there preoperatively, and transferred back to the same ward postoperatively for further treatment and rehabilitation, while the control group will be treated in a traditional orthopaedic ward. Operative and anaesthesiologic procedures will be the same in the two groups.

The primary endpoint is chosen in order to optimize clinical relevance as well as sensitivity to change within a wide range of functional performance, and will be recorded four months after the fracture. Our main hypothesis is that an orthogeriatric service may improve long-time cognitive outcome. Accordingly, we will use a composite endpoint tapping cognitive functioning in the lower as well as the higher spectre of performance by these two instruments:

* Clinical Dementia Rating Scale (CDR), proxy-based scale for severity of dementia, that is able to detect differences also between patients with severe dementia. The scale consists of six questions, each rated 0-3, adding up to a sumscore of 0-18 ("sum of boxes"). The scale is frequently used in dementia treatment trials, and is shown to be valid and reliable. CDR will be scored based on the best available source (relative, staff in nursing home or home nursing service)
* The 10 words memory task from the Consortium to Establish a Registry for Alzheimer's Disease battery (CERAD). This test is shown to be sensitive for memory changes in persons that have a good or fairly good cognitive functioning. We will use the immediate recall and the delayed recall parts of this task, i.e. two scales.

The primary endpoint will be assessed after four months, by a specially trained research assistant blinded to allocation. The patients will be re-assessed after 12 months.

ELIGIBILITY:
Inclusion Criteria:

• Eligible patients will be admitted acutely for a femoral neck fracture, a trochanteric or a subtrochanteric femoral fracture.

Exclusion Criteria:

* Hip fracture as part of multi-trauma or high energy trauma (defined as a fall from a higher level than 1 metre). One recent fracture in addition to the hip fracture (e.g. radius or shoulder) is acceptable.
* Regarded as moribund at admittance.
* Absence of a valid informed consent or assent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
We will use a composite endpoint by these two instruments: Clinical Dementia Rating Scale (CDR), and the 10 words memory task from the Consortium to Establish a Registry for Alzheimer's Disease battery (CERAD) | 4 and 12 months

SECONDARY OUTCOMES:
Activities of Daily Living (ADL) Scale | 4 and 12 months
Nottingham Extended Activities of Daily Living (NEADL) scale | 4 and 12 months
Intrahospital mortality | 4 and 12 months
Cumulative mortality | 4 and 12 months
The Short Physical Performance Battery (SPPB) scale | 4 and 12 months
Pre-/postoperative delirium | 4 and 12 months
Duration/Severity of delirium | 4 and 12 months
Other complications | 4 and 12 months
Incidence of dementia 12 months postoperatively | 4 and 12 months
Length of hospital stay | 4 and 12 months
Markers of bone turnover | 4 months
Micronutrients in blood | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Bruun Wyller, MD, Prof., Study Director — University of Oslo, Fac of Med., Geriatric dep.
Locations (1):
- Oslo University Hospital, Ullevaal, Oslo, Norway

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Torbergsen AC, Watne LO, Frihagen F, Wyller TB, Mowe M. Effects of nutritional intervention upon bone turnover in elderly hip fracture patients. Randomized controlled trial. Clin Nutr ESPEN. 2019 Feb;29:52-58. doi: 10.1016/j.clnesp.2017.11.012. Epub 2018 Oct 30. PMID 30661701
- [Derived] Torbergsen AC, Watne LO, Wyller TB, Frihagen F, Stromsoe K, Bohmer T, Mowe M. Micronutrients and the risk of hip fracture: Case-control study. Clin Nutr. 2017 Apr;36(2):438-443. doi: 10.1016/j.clnu.2015.12.014. Epub 2015 Dec 23. PMID 26795217
- [Derived] Watne LO, Torbergsen AC, Conroy S, Engedal K, Frihagen F, Hjorthaug GA, Juliebo V, Raeder J, Saltvedt I, Skovlund E, Wyller TB. The effect of a pre- and postoperative orthogeriatric service on cognitive function in patients with hip fracture: randomized controlled trial (Oslo Orthogeriatric Trial). BMC Med. 2014 Apr 15;12:63. doi: 10.1186/1741-7015-12-63. PMID 24735588
- [Derived] Wyller TB, Watne LO, Torbergsen A, Engedal K, Frihagen F, Juliebo V, Saltvedt I, Skovlund E, Raeder J, Conroy S. The effect of a pre- and post-operative orthogeriatric service on cognitive function in patients with hip fracture. The protocol of the Oslo Orthogeriatrics Trial. BMC Geriatr. 2012 Jul 20;12:36. doi: 10.1186/1471-2318-12-36. PMID 22817102